CLINICAL TRIAL: NCT05702502
Title: Liquid Biopsy for the Identification of Malignancy Associated Haemophagocytic Lymphohistiocytosis (HLH)
Brief Title: Assessing the Presence of CT-DNA in Lymphoma Associated HLH
Status: Recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22CH022
Record Dates: First submitted 2022-09-28; First posted 2023-01-27 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma; Haemophagocytic Lymphohistiocytosis
MeSH Terms: conditions — Lymphoma; Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating tumour DNA Tumour biopsy Peripheral blood white cells (for germline DNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Haemophagocytic lymphohistiocytosis (HLH) is a rare life-threatening blood disease which causes severe inflammation with symptoms similar to severe sepsis. It is hard to diagnose. The most common cause of HLH in adults is lymphoma (blood cancer). Outcomes for adults with HLH and cancer are serious, and most die after days or weeks because they have been diagnosed or treated too late. It is likely that many cases where patients died of HLH with no underlying cause actually had cancer.

Recently it has been found that patients with certain types of lymphoma have DNA which comes directly from their cancer (circulating tumour DNA; ctDNA). Aggressive lymphomas release a lot of ctDNA which can be detected in the blood of patients. This study will look for ctDNA in patients with HLH, and see if it is possible to use it to diagnose lymphoma earlier. Patients will provide a small additional blood sample for analysis. Diagnosing lymphoma more rapidly would mean more people could get the correct treatment for the lymphoma which has caused their HLH. They could receive the correct treatment sooner. Earlier diagnosis and treatment could improve survival for these patients.

DETAILED DESCRIPTION:
A variety of constitutive and acquired risks trigger HLH. In general, infants have inherited T- and NK-cell defects impairing cytotoxic function, while adults are most likely to suffer from lymphoma, most commonly diffuse large B cell lymphoma (DLBCL), Hodgkin lymphoma and T-cell lymphoma. Patients with underlying lymphoma have the worst survival rates (West et al J Intern Med 2021). Diagnosis of lymphoma is challenging due to severe sepsis-like presentation, meaning CT-PET and early biopsy may not be possible. Patients with delayed/no diagnosis frequently receive empirical chemotherapy, delaying diagnosis, inadequately treating underlying lymphoma and potentially worsening infections. Epidemiological studies have failed to show improvements in survival in patients with HLH, whilst also confirming a significant increase in the number of diagnoses (West et al J Intern Med 2021). Improvements in rapidly diagnosing cases of lymphoma driving HLH would result in better outcomes due more rapid (immuno-)chemotherapy administration.

Circulating tumour DNA (ctDNA) are DNA isolated from blood, originating from the apoptosis/necrosis of cancerous cells. ctDNA reflects the entire tumour genome and is referred to as a "liquid biopsy". These techniques are under investigation in several lymphomas, and DLBCL-specific mutations can be detected and quantified using ctDNA, with studies using quantification as a strategy to monitor response to therapy (Kurtz et al J Clin Onc 2018). Similarly, ctDNA mutations can be identified in Hodgkin lymphoma (Spina et al Blood 2018) and T-cell lymphoma (Ottolini et al Blood advances 2020).

Capitalising on the success of the DLBCL Interim Response Evaluation for Customised Therapy (DIRECT) study, existing infrastructure in Cambridge will be used to conduct a feasibility study assessing whether ctDNA from patients with HLH with underlying lymphoma is viable in contributing to diagnoses. Blood samples from patients with HLH will have ctDNA and granulocytes extracted and stored. Once lymphoma is confirmed, the biopsy will be requested and ctDNA, granulocytes and biopsy from each patient will be interrogated using shallow whole genome sequencing (WGS; 0.1x) and a high-sensitivity, targeted sequencing panel termed LyVE-Seq (~2000x). This panel includes coding regions of 122 genes implicated as drivers of DLBCL, in addition to translocation hotspots for BCL6/MYC. For non-DLBCL, the existing panel will be modified to include 150 genes recurrently mutated across all lymphoma subtypes, ordered as a focused panel from Twist Bioscience.

Demographic/laboratory data will be requested and will be integrated with information from clinical risk scores, tumour genotype, and radiology (CT/PET-CT). These invaluable clinical samples will be stored and may be used for future research as, to date, there is no data for ctDNA in the context of malignancy associated HLH and the study is highly exploratory.

ELIGIBILITY:
Inclusion criteria:

* Informed consent.
* Age ≥18 years.
* Clinically confirmed HLH.
* High dose steroids and/or systemic anti-cancer therapy (SACT) for <72 hours for the current episode of HLH (anakinra is not considered SACT). Prior steroid use >14 days at the time of consent is permitted.
* Patients with recurrent HLH may be included.
* Patients already known to have underlying lymphoma, or have relapsed lymphoma may be included.

Exclusion criteria:

• Cause of HLH already known to be due to a non-malignant cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HLH are usually unwell and hospitalised. Patients will be identified by the clinical (direct care) teams following a clinical diagnosis of HLH as part of routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Identification of lymphoma-specific mutations in ctDNA from patients with lymphoma driven HLH. | Up to 2 years
  For those patients found to have lymphoma driven haemophagocytic syndrome we will assess whether we can find the presence of cell free tumour DNA in blood.

SECONDARY OUTCOMES:
Assess the utility of integrated data from clinical risk factors (IPI), up-front genotype, and radiological assessment (CT or PET-CT) with ctDNA findings. | Up to 2 years
  We will use clinical, radiological and tumour mutation status to see if there is any correlation with the detection of cell free tumour DNA.
Assessing the feasibility of returning central laboratory data in a clinically useful timeframe. | Up to 2 years
  Provided the primary outcome is successful we will see if the finding of cell free tumour DNA can be used as a clinical test to identify lymphoma in patients with HLH,

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Univeristy Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom